CLINICAL TRIAL: NCT00176358
Title: Percutaneous Coronary Angioplasty Compared With Exercise Training in Symptomatic Coronary Artery Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139/2001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-09-10 (Estimated); Status verified 2005-09

CONDITIONS: CAD; Stable Angina Pectoris
MeSH Terms: conditions — Angina, Stable | interventions — Exercise

INTERVENTIONS:
Device: PTCA and Stent Implantation
Behavioral: Exercise Training

SUMMARY:
The purpose of this study is to compare coronary angioplasty with stent implantation with an exercise rehabilitation program in patients with stable coronary artery disease (CAD).

ELIGIBILITY:
Inclusion Criteria:

* Angiographically documented CAD, with at least one coronary artery stenosis of more than 50% in a native segment never subjected to intervention, which is recommended for treatment with percutaneous transluminal coronary angioplasty (PTCA).
* Stable coronary artery disease
* Eligible patients could be asymptomatic or have class I to III angina (Canadian Cardiovascular Society [CCS]) with documented myocardial ischemia
* Angina pectoris threshold > 50 Watt (cycle ergometry)
* Permanent residence should be within 25 km of training facility.

Exclusion Criteria:

* < 18 or > 70 years of age
* Patient currently participating in an exercise training program
* Unstable angina pectoris or myocardial infarction during the last 2 weeks
* Symptoms of CCS class IV
* Exercise limitations due to clinical conditions not related to CAD
* Left ventricular ejection fraction (LVEF) of < 40%
* Ventricular arrhythmia (Lown Ivb)
* Hemodynamically significant valvular heart disease
* Previous cardiac surgery
* PTCA performed during the last 12 months
* Any major non-cardiac condition that would adversely affect survival during the duration of the study
* Reduced compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Hambrecht, Prof., Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany